CLINICAL TRIAL: NCT01486277
Title: A Phase 2, Single-arm, Open-label, Multicenter Study of the Histone Deacetylase Inhibitor (HDACi) JNJ-26481585 in Subjects With Previously Treated Stage Ib-IVa Cutaneous T-cell Lymphoma
Brief Title: A Study of the Histone Deacetylase Inhibitor (HDACi) Quisinostat (JNJ-26481585) in Patients With Previously Treated Stage Ib-IVa Cutaneous T-cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR018640; 2011-001076-18 (EudraCT Number); 26481585LYM2001 (Other: Janssen Research & Development, LLC); NCT01389960 (obsolete NCT alias)
Record Dates: First submitted 2011-11-29; First posted 2011-12-06 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Lymphoma, T-Cell, Cutaneous
Keywords: Lymphoma, T-Cell, Cutaneous; T-cell lymphoma; Lymphoma; Histone Deacetylase Inhibitor; JNJ-26481585
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Lymphoma, T-Cell; Lymphoma | interventions — quisinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Quisinostat (Experimental): Participants will receive quisinostat 12 mg capsule orally (by mouth) on Days 1, 3, and 5 of each week in a 21-day treatment cycle, until a reason for discontinuation is met (ie, disease progression, toxicity, availability of other effective medications that the participant may receive, or treating physician advice).
  Interventions: Drug: Quisinostat, 12 mg

INTERVENTIONS:
Drug: Quisinostat, 12 mg — Participants will receive quisinostat 12 mg capsule orally (by mouth) on Days 1, 3, and 5 of each week in a 21-day treatment cycle, until a reason for discontinuation is met (ie, disease progression, toxicity, availability of other effective medications that the participant may receive, or treating physician advice).
  Other Names: JNJ 26481585

SUMMARY:
The purpose of this study is to determine the overall cutaneous response rate (participants who achieve a complete response or partial response) based on the modified severity weighted assessment tool criteria.

DETAILED DESCRIPTION:
This is a single-arm (group), open-label (all people know the identity of the intervention), and multicenter study. The study consists of 3 phases including, the screening phase (within 28 days prior to the start of study medication), treatment phase (participants will receive quisinostat) and follow-up phase (30 days after the last dose of study medication until death or clinical cutoff). Clinical cut-off is defined as when the last participant will be assessed with progressive disease or died, or 6 months after the last participant enrolled, whichever occurs first. However, if any participants are still receiving study treatment at the time of clinical cut-off, these participants will enter a long-term extension phase and will continue to receive study medication until a reason for discontinuation is met (ie, disease progression, toxicity, availability of other effective medications that the participant may receive, or treating physician advice). The long-term extension phase will continue for a maximum of 2 years beyond the clinical cut-off for primary analysis. Safety will be evaluated by the assessment of adverse events, vital signs, physical examination, 12-lead electrocardiogram, and clinical laboratory tests which will be monitored in this study. Any participants responding to treatment at the end of the 2-year long-term extension phase will be able to continue to receive quisinostat as long as they are assessed by the investigator as not meeting treatment discontinuation criteria; during this time, only information related to serious adverse events will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed cutaneous T-cell lymphoma (CTCL), either mycosis fungoides or sezary syndrome Stage Ib-IVa
* Relapsed or refractory (unresponsive) disease following at least 1 prior systemic therapy for CTCL, except psoralen and long-wave ultraviolet radiation (it is considered skin-directed therapy and not systemic therapy)
* Stable anti-pruritus regimen (topical corticosteroids or antihistamine) in the preceding 28 days
* Measurable disease with at least 1 skin lesion (patch, plaque, or tumor) 1 cm or greater than 1 cm in the longest diameter laboratory function tests and bone marrow test
* Agrees to protocol defined use of effective contraception
* Adequate laboratory function tests and bone marrow test

Exclusion Criteria:

* Prior histone-deacetylase inhibitor therapy for CTCL
* Concurrent systemic corticosteroid dose greater than 10 mg per day of prednisone or equivalent (stable use of 10 mg or less than 10 mg per day of prednisone for 1 month or more before study entry is allowed)
* Major surgery or radiotherapy within 3 weeks before the start of the study medication
* Unstable angina or heart attack within the preceding 12 months, congestive heart failure New York Heart Association Class II-IV, known presence of dilated, hypertrophic, or restrictive cardiomyopathy
* Inadequate gastrointestinal absorption status
* Use of potent inhibitors of CYP3A4/A5
* Positive human immunodeficiency virus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-11; Primary Completion 2014-11 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Number of participants who will achieve overall cutaneous Response Rate (RR) based on modified Severity Weighted Assessment Tool (mSWAT) criteria | From screening until progressive disease or confirmed lost to follow-up or death or start of alternate therapy, or withdrawal from the study; as assessed for approximately 6 months after the enrollment of the last participant
  The RR is defined as the number of participants who will achieve a complete response (CR) or partial response (PR). mSWAT criteria is used to evaluate the skin tumor burden. The investigator will determine the percentage of total body surface area (TBSA) affected by patches, plaques or tumors in 12 body regions, using the participant's palm and fingers representing 1% of TBSA. CR is defined as 100% clearance of skin lesions and PR is defined as 50% to 99 % clearance of skin lesions from baseline without occurrence of a new tumor.

SECONDARY OUTCOMES:
Number of participants who will achieve global Response Rate (RR) based on based on consensus global response score | From screening until progressive disease or confirmed lost to follow-up or death from any cause or start of alternate therapy, or withdrawal from the study; as assessed for approximately 6 months after the enrollment of the last participant
  The RR is defined as the number of participants who will achieve a complete response (CR) or partial response (PR). Global response score provides uniformity in the assessment of response and utilizes all component of the tumor-node-metastasis-blood staging (ie, skin, nodes, viscera and blood). Complete response is defined as complete disappearance of all clinical evidence of disease (all categories have CR/ non-involved [NI]) and PR is defined as regression of measurable disease (all categories do not have a CR/NI and no category has a PD and if any other category involved at baseline, at least one has a CR or PR).
Progression-Free Survival (PFS) | From the date of administration of the first dose of study medication until progressive disease or death from any cause, whichever occurs first; as assessed for approximately 6 months after the enrollment of the last participant
  PFS is defined as the interval between the date of administration of the first dose of study medication and the date of disease progression or death from any cause, whichever occurs first.
Kaplan-Meier Estimates of 1-year overall survival (OS) rate | From the date of administration of the first dose of study medication up to the date of progressive disease or death, whichever occurs first; as assessed up to 1 year
  1-year OS rate is defined as the number of participants surviving at 1 year after the date of administration of the first dose of study medication.
Duration of response (DOR) for participants achieving Complete Response (CR) or Partial Response (PR) | First documentation of CR or PR until the date of first documentation of progressive disease, or death from any cause; as assessed for approximately 6 months after the enrollment of the last participant
  DOR for participants achieving a CR or PR is defined as the date from the first documentation of CR or PR until the date of first documentation of progressive disease, or death from any cause.
The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | From screening until progressive disease or confirmed lost to follow-up or death from any cause or start of alternate therapy, or withdrawal from the study; as assessed for approximately 6 months after the enrollment of the last participant
  EORTC QLQ-C30 is a questionnaire to assess quality of life of cancer patients. It is composed of 30 items, multi-item measure (28 items) and 2 single-item measures. For the multiple item measure, 4-point scale is used and the score for each item range from "1 = not at all" to "4 = very much". Higher scores indicate worsening. The 2 single-item measure involves question about the overall health and overall quality of life which will be rated on a 7-point scale ranging from "1 = very poor" to "7 = excellent". Lower scores indicate worsening.
Pruritus Intensity Assessment Questionnaire scale scores | From screening until progressive disease or confirmed lost to follow-up or death from any cause or start of alternate therapy, or withdrawal from the study; as assessed for approximately 6 months after the enrollment of the last participant
  Pruritus Intensity Assessment Questionnaire is an 11-point scale that requires the participant to rate the intensity of their pruritus. The scores range from '0= no pruritus; 10 = worst imaginable'. Pruritus relief will be defined as a 3 or more point decrease in participant who have a baseline pruritus score of 3 or more points or complete resolution of pruritus for 3 or more continuous weeks without an increase in the use of antipruritic medications. Higher score indicates worsening.
Number of participants with adverse events | Up to 2 years after 6 months enrollment of the last participant

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (13):
- Pittsburgh, Pennsylvania, United States
- France (3):
  - Nantes
  - Paris
  - Pessac
- Germany (2):
  - Kiel
  - Minden
- Portugal (2):
  - Lisbon
  - Porto
- Spain (3):
  - Madrid
  - Málaga
  - Valencia
- United Kingdom (2):
  - London
  - Manchester